CLINICAL TRIAL: NCT00051766
Title: A Computer-Based HIV Medication Adherence Intervention
Brief Title: Computer-Assisted Adherence Program for Patients Taking Anti-HIV Drugs
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: 2R44AI044558-02A1 (NIH)
Record Dates: First submitted 2003-01-16; First posted 2003-01-17 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2005-05

CONDITIONS: Acquired Immunodeficiency Syndrome; HIV Infections
Keywords: compliance; medication; antiretroviral; adherence; intervention; treatment experienced
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections; Patient Compliance

INTERVENTIONS:
Behavioral: Computer-based Intervention

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a computer-assisted, self-administered adherence program for patients on complicated anti-HIV drug regimens.

DETAILED DESCRIPTION:
Highly active antiretroviral therapy (HAART) for HIV produces dramatic reductions in morbidity and mortality for many patients who maintain a high level of adherence to their medications. However, 20% to 33% of HIV infected patients will miss at least one of their medication doses over a one to three day period. Patient self-report is the most practical method for assessing adherence, but it may produce unreliable and invalid results unless optimally performed. A computer-assisted, self-administered adherence program could improve HIV infected patients' adherence behaviors by accurately and efficiently assessing their medication adherence, delivering an adherence intervention to patients, and producing adherence reports for providers. By providing a neutral and seemingly private interview, computer programs may increase patient disclosure of non-adherence. This study will evaluate the efficacy of a computer-assisted, self-administered adherence program in reducing regimen misunderstandings and enhancing patient adherence.

Participants in this study will be recruited from within the Positive Health Program at San Francisco General Hospital. Patients will be randomly assigned to a Control or Intervention Group. Control Group participants will complete an audio computer-assisted self-interview (A-CASI) assessing their understanding of their medication regimen and adherence. Intervention Group participants will complete the adherence A-CASI and will receive a brief computer-delivered intervention consisting of a graphical depiction of their correct regimen and strategies for improving adherence. Study investigators will forward a computer-generated adherence report, which summarizes their adherence and suggests appropriate interventions, to the Intervention Group's health care providers. All participants will be assessed at least three times over a 6-month period: study entry, Month 3, and Month 6.

ELIGIBILITY:
Inclusion Criteria

* Receiving HIV care at San Francisco General Hospital's Positive Health Program
* Three or more antiretroviral medications
* HIV-1 viral load > 500 copies/ml
* At least one previous salvage regimen
* Ability to read English at 8th grade level

Exclusion Criteria

* Visual impairments that prevent patient from reading text on a computer screen
* Obvious cognitive impairment

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200

CONTACTS AND LOCATIONS:
Overall Officials: Frederick M. Hecht, MD, Study Chair — San Francisco General Hospital; Amy B. Bronstone, PhD, Study Director — West Portal Software Corporation; Roger Hofmann, BS, Principal Investigator — West Portal Software Corporation
Locations (1):
- San Francisco General Hospital, San Francisco, California, United States